CLINICAL TRIAL: NCT06834581
Title: Effects of Vibrating Mesh Nebulisation in Patients on Long-term Tracheostomy Ventilation: a Pilot Randomised Crossover Trial
Acronym: EVOLVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 348268
Record Dates: First submitted 2025-02-06; First posted 2025-02-19 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Long-term Tracheostomy Ventilated Patients
Keywords: vibrating mesh nebuliser; jet nebuliser; long-term tracheostomy ventilated patients

STUDY DESIGN:
Intervention Model Description: Pilot randomised crossover trial
Who Masked: Outcomes Assessor
Masking Description: VMN and JN are easily distinguishable due to both their visible and audible signatures. It is therefore not feasible to blind the patient to the delivered intervention. The mode of nebulisation will be known to both the investigator and participant, and the absence of masking is acknowledged to be a potential source of bias. NRD and spirometry analysis will be masked as off-line analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vibrating mesh nebulisation then jet nebulisation (Experimental): Participants will receive hypertonic saline and salbutamol via vibrating mesh nebulisation for the first 30 hours. After a 24-hour washout period, they will receive the same medications via jet nebulisation.
  Interventions: Device: Vibrating mesh nebuliser; Device: Jet nebuliser
- Jet nebulisation then vibrating mesh nebulisation (Experimental): Participants will receive hypertonic saline and salbutamol via jet nebulisation for the first 30 hours. After a 24-hour washout period, they will receive the same medications via vibrating mesh nebulisation.
  Interventions: Device: Vibrating mesh nebuliser; Device: Jet nebuliser

INTERVENTIONS:
Device: Vibrating mesh nebuliser — Vibrating mesh nebulisation (VMN) uses a mesh membrane that oscillates at high frequency (typically 128 kHz) to produce a stream of drug-carrying droplets of pre-determined size to be inhaled.
Device: Jet nebuliser — Jet nebulisers use the flow of a gas (air or oxygen) to draw medication up through a capillary tube to generate small particles to be inhaled.

SUMMARY:
Assessment of the effects of vibrating mesh nebulisation versus jet nebulisation on respiratory function in patients with long-term tracheostomy ventilation: evaluating neural respiratory drive, breathing mechanics, cardiac parameters, secretions, and breathlessness

DETAILED DESCRIPTION:
Long-term tracheostomy ventilation (LTTV) is frequently complicated by high secretion burden, arising from accumulation of oronasal and bronchial secretions due to impaired bulbar or cough function. Patients are therefore at an increased risk of sputum plugging and respiratory infection, leading to potentially life-threatening deterioration. In patients undergoing weaning from prolonged mechanical ventilation, liberation from invasive mechanical ventilation can be delayed by excessive secretion burden, detrimentally affecting quality of life and escalating healthcare costs.

The principal treatment strategies for secretion retention are oral and tracheal suction, mucolytic therapy (enteral or nebulised) and mechanical insufflation-exsufflation (MIE). There are few robust data to support the use of these treatment modalities, although they are routinely used in clinical practice on an empirical basis. The use of nebulised hypertonic saline is well-established in the management of non-cystic fibrosis bronchiectasis and is frequently used to aid airway clearance in LTTV patients. Nebulised salbutamol is widely used as a bronchodilator in tracheostomised patients with a tendency to develop bronchospasm, whether due to established obstructive airways disease or airways inflammation from secretion retention or ventilator-associated pneumonia.

Vibrating mesh nebulisation (VMN) is increasingly used for aerosol delivery in mechanically ventilated patients, with advantages including reduced residual volume, quieter operation and higher levels of drug deposition. However, its superiority in improving secretion clearance and bronchodilation compared with jet nebulisation (JN) is yet to be established. Both VMN and JN are currently utilised within clinical practice as standards of care.

This pilot randomised crossover trial seeks to recruit 12 patients to establish whether VMN of hypertonic saline and salbutamol has a greater effect than standard JN in improving:

Neural respiratory drive (measured by assessment of the electrical activity of breathing muscles via parasternal EMG) Secretion burden Breathlessness

Participants will be recruited as inpatients within the Lane Fox Unit. Following consent for trial involvement, there will be a 24-hour washout period receiving normal saline nebulisers. Baseline data including ventilator settings, anthropometrics and clinical observations will be recorded before participants are randomly allocated to receive salbutamol and hypertonic (3%) saline via either VMN or JN four times per day for 30 hours. During this period, measurements will include:

Neural respiratory drive (via parasternal EMG) Carbon dioxide levels (via forehead probe) Breathlessness and sputum burden (using numerical scales) 24-hour sputum volume with samples for bacterial/viral analyses

Following a 24-hour washout period, participants will receive salbutamol and hypertonic saline via the alternative nebuliser type for 30 hours, with identical data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving long-term tracheostomy ventilation as inpatients of the Lane Fox Respiratory Service at Guy's and St Thomas' NHS Foundation Trust
* Requiring prolonged mechanical ventilation for at least 6 hours per day for at least 21 days
* Has a cuffed tracheostomy in situ
* Aged 18-80 years old
* Receiving normal (0.9%) saline or hypertonic saline nebulisation at the time of enrolment into the study
* Requiring and tolerating tracheal suctioning for secretion management
* Able to communicate symptom burden to the research team
* Able to give informed consent for participation in the study
* Clinical stability, with no requirement for changes in ventilatory support, as assessed by the responsible clinician for at least 48 hours prior to enrolment in study

Exclusion Criteria:

* Severe, non-respiratory organ dysfunction including, but not limited to:

  * Congestive cardiac failure
  * Cardiac arrhythmia
  * End-stage malignancy
  * End-stage renal failure
* Acute pulmonary pathology requiring emergency treatment including, but not limited to:

  * Ventilator associated pneumonia at the time of screening
  * Pneumothorax
  * Pulmonary embolism
* Severe cognitive impairment
* Psychosocial factors that would preclude completion of the study protocol
* Previous intolerance of aerosolised hypertonic 3% saline or nebulised salbutamol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Neural Respiratory Drive | At baseline and during both 30 hour nebuliser allocations. Following nebulisation measurements to be made at 15 and 30 minutes
  Parasternal electromyography, which reflects the load-capacity relationship of the respiratory system, will likely decrease with more effective bronchodilation and secretion clearance.

SECONDARY OUTCOMES:
Sputum viscosity | Daily during both 30 hour periods
  Sputum viscosity will be measured by a single assessor using the Qualitative Sputum Analysis Tool (QSAT) score daily during both 30-hour periods. The QSAT score includes sputum volume, type (mucoid, mucopurulent and purulent) and grades viscosity from 1 (adherent) to 4 (easily pourable) in 0.5 increments.
Sputum weight | At baseline and during both 30 hour nebuliser periods
  24 hour cumulative wet sputum weight will be measured at baseline and during each nebuliser phase
Heart rate | At baseline and during 2 x 30 hour periods
  Heart rate will be assessed by continuous ECG monitoring to detect changes following administration of salbutamol and hypertonic saline by VMN versus JN. Heart rate will be measured in beats per minute.
Respiratory Flow | At baseline and during each 30 hour time period
  Assessment of respiratory flow via pneumotach within both 30 hour time periods
Symptoms of breathlessness (modified Borg dyspnea scale) | At baseline and during both 30 hour nebulisation periods
  Patient perception of breathlessness will be assessed using the modified Borg dyspnoea scale (mBorg). The scale ranges from 0 to 10 (whole numbers plus 0.5), where 0 indicates no breathing difficulty and 10 represents maximal breathing difficulty.
Symptoms of breathlessness (numerical rating scale) | At baseline and during both 30 hour nebulisation periods
  Patient perception of breathlessness will be assessed using a numerical rating scale from 0 to 10, where 0 represents no breathlessness and 10 represents the worst breathlessness imaginable.
Symptoms of sputum burden | At baseline and during both 30 hour nebulization periods
  Patient perception of secretion burden will be assessed using a numerical rating scale rated from 0 to 10, where 0 represents no burdensome secretions and 10 represents secretions being the worst imaginable.
Heart Rhythm | At baseline and during the 2 x 30 hour periods
  Changes in heart rhythm will be assessed by ECG monitoring to detect variations following administration of salbutamol and hypertonic saline by VMN versus JN. Any changes in heart rhythm or arrhythmias will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Eui Sik Suh, MBBS MChem(Oxon) PhD FRCP, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Lane Fox Unit, St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnott A, Hart R, McQueen S, Watson M, Sim M. Prospective randomised unblinded comparison of sputum viscosity for three methods of saline nebulisation in mechanically ventilated patients: A pilot study protocol. PLoS One. 2023 Aug 17;18(8):e0290033. doi: 10.1371/journal.pone.0290033. eCollection 2023. PMID 37590203
- [Background] Kellett F, Redfern J, Niven RM. Evaluation of nebulised hypertonic saline (7%) as an adjunct to physiotherapy in patients with stable bronchiectasis. Respir Med. 2005 Jan;99(1):27-31. doi: 10.1016/j.rmed.2004.05.006. PMID 15672845
- [Background] Tarrant BJ, Le Maitre C, Romero L, Steward R, Button BM, Thompson BR, Holland AE. Mucoactive agents for chronic, non-cystic fibrosis lung disease: A systematic review and meta-analysis. Respirology. 2017 Aug;22(6):1084-1092. doi: 10.1111/resp.13047. Epub 2017 Apr 11. PMID 28397992
- [Background] Anand R, McAuley DF, Blackwood B, Yap C, ONeill B, Connolly B, Borthwick M, Shyamsundar M, Warburton J, Meenen DV, Paulus F, Schultz MJ, Dark P, Bradley JM. Mucoactive agents for acute respiratory failure in the critically ill: a systematic review and meta-analysis. Thorax. 2020 Aug;75(8):623-631. doi: 10.1136/thoraxjnl-2019-214355. Epub 2020 Jun 8. PMID 32513777
- [Background] Mifsud Bonnici D, Sanctuary T, Warren A, Murphy PB, Steier J, Marino P, Pattani H, Creagh-Brown BC, Hart N. Prospective observational cohort study of patients with weaning failure admitted to a specialist weaning, rehabilitation and home mechanical ventilation centre. BMJ Open. 2016 Mar 8;6(3):e010025. doi: 10.1136/bmjopen-2015-010025. PMID 26956162